CLINICAL TRIAL: NCT04131413
Title: A Phase I Open Label, Dose Escalation Clinical Trial Assessing the Safety, Tolerability, and Feasibility of pNGVL4aCRTE6E7L2 HPV DNA Vaccine Administration Via Intramuscular TriGridTM Electroporation Delivery System to Patients With HPV16-Positive High-Grade Cervical Intraepithelial Neoplasia
Brief Title: HPV DNA Vaccine Via Electroporation for HPV16 Positive Cervical Neoplasia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J1955; IRB00197468 (Other: Johns Hopkins University Institutional Review Board); 118209 (Other: National Cancer Institute)
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Human Papillomavirus Type 16; Cervical Intraepithelial Neoplasia Grade II; Cervical Intraepithelial Neoplasia, Grade III
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: Three dose level cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vaccination Arm Level 1 (Other): The dose escalation of pNGVL4aCRTE6E7L2 will be conducted to evaluate the safety of three escalating doses; Level 1 dose of 0.3 mg
  Interventions: Drug: pNGVL4aCRTE6E7L2
- Vaccination Arm Level 2 (Other): The dose escalation of pNGVL4aCRTE6E7L2 will be conducted to evaluate the safety of three escalating doses; level 2 at dose 1.0 mg
  Interventions: Drug: pNGVL4aCRTE6E7L2
- Vaccination Arm Level 3 (Other): The dose escalation of pNGVL4aCRTE6E7L2 will be conducted to evaluate the safety of three escalating doses; level 3 dose of 3.0 mg
  Interventions: Drug: pNGVL4aCRTE6E7L2

INTERVENTIONS:
Drug: pNGVL4aCRTE6E7L2 — The dose escalation will start from the lowest dose level of 0.3 mg. This dose cohort will consist of 3 participants and a monitoring period of one week after the final dose mandated. If there are 0 participants in the 0.3 dose level cohort that experience dose limiting toxicities (DLT), a new cohort of 3 participants will be vaccinated at the 1.0 mg dose level. If there are 0 participants in the 1.0 mg dose level that experience DLT, then a new cohort of 3 participants will be vaccinated at the 3.0 mg dose level. If there is 1 participant experiencing DLTs, an additional cohort of 3 subjects will be enrolled and treated at the current dose level. If there are 2 or more participants experiencing DLTs in the 3 or additional cohort of 3 vaccinated at the current dose level, then the next lower dose level will be determined as the Maximum Tolerated Dose (MTD).

SUMMARY:
The primary goal of this phase I open label study is to determine the safety and tolerability of pNGVL4aCRTE6E7L2 DNA vaccine, as administered by intramuscular (IM) injection with TriGrid™ electroporation to both HIV- or HIV+ adult female subjects (≥ 19 years), with biopsy confirmed cervical intraepithelial (CIN) II or III that is human papillomavirus (HPV) 16+.

ELIGIBILITY:
Inclusion Criteria:

* For the HIV- patient cohort only: patients with high-grade cervical intraepithelial lesions (CIN2/3) confirmed by colposcopy and biopsy who are HIV negative
* For the HIV+ patient cohort only: patients with high-grade cervical intraepithelial lesions (CIN2/3) confirmed by colposcopy and biopsy that are HIV positive

  1. HIV-1 infection, as documented by a rapid HIV-1 test or any FDA-approved HIV-1 enzyme or chemiluminescence immunoassay (E/CIA) test kit and confirmed by western blot at any time prior to study entry.
  2. Two HIV-1 RNA values ≤200 copies/mL at least 24 hours apart performed by any laboratory that has Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent may be used to document infection.
  3. Patients must be willing to comply with effective Antiretroviral Therapy.
* Patients whose cervical cytologic samples are HPV16+ by Roche Cobas 4800, Roche Linear Array HPV Genotyping test or other FDA-approved HPV genotyping test. Co-infections with HPV types other than HPV16 are permissible for study entry.
* Age ≥19 years. Also due to Alabama law the age a person is no longer a minor needing parental consent is 19, so all participants need to be 19 or older.
* Life expectancy of greater than 4 months.
* Baseline Eastern Cooperative Oncology Group performance status of 0, 1 at the time of multi-modality treatment administration
* Participants must have normal organ and marrow function within 45 days of enrollment as defined below:

Absolute neutrophil count > 1,500/mcL Cluster of differentiation (CD) 4 cell count > 200/mcL Platelets > 100,000/mcL Hemoglobin > 10.0 g/dL Total bilirubin < 1.5 X upper institutional limit of normal (patients with diagnosed Gilbert's Syndrome will not be excluded if direct bilirubin is within normal institutional limits) aspartate aminotransferase (AST) <1.5 X the upper institutional limit of normal Alanine transaminase (ALT) <1.5 X the upper institutional limit of normal Creatinine ≤1.5 x upper institutional limit normal

* The effects of pNGVL4aCRTE6E7L2 DNA vaccine on the developing human fetus is unknown. For this reason, women of child-bearing potential must agree to use two forms of acceptable contraception, including one barrier method, prior to study entry and for 3 months after study completion. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.

  1. Women of childbearing potential are defined as any female who has experienced menarche and does not meet the criteria for "women not of childbearing potential" defined below.
  2. Women not of childbearing potential are defined as follows:

  i. Women who are permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) ii. Women who have experienced total cessation of menses for at least 1 year OR who have a previous clinical follicle stimulating hormone (FSH) value > 40 mIU/mL c. The following are acceptable forms of barrier contraception: i. Male or female condom, ii. Diaphragm, cervical/vault cap, or contraceptive sponge when used with spermicidal foam/gel/cream/suppository.

  d. The following are acceptable forms of secondary contraception, when used with a barrier method and spermicide: i. Placement of an intrauterine device (IUD) ii. Established use of oral, injected, or implanted hormonal methods of contraception
* Ability to understand and the willingness to sign a written informed consent document.
* Participant is able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Patients with high-grade cervical intraepithelial lesions (CIN2/3) that are HPV16 negative
* For the HIV+ cohort only: patients with AIDS related symptoms comprising an active AIDS-associated infectious process that, in the view of the investigator, would limit the subject's ability to comply with study procedures.
* For the HIV+ cohort only: patients with an HIV viral load >200 cp/mL.
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within 6 months of study entry; For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day; inhaled and topical steroids are allowed.
* Due to interference with the immunologic measurements and compromising the analysis of the safety of the vaccine, participants with active or chronic infection of hepatitis C virus (HCV) or hepatitis B virus (HBV) are excluded as well as those who have previously received an investigational HPV vaccine.
* Participants who are receiving or have received any other investigational agents within 30 days of registration.
* Participants with an uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic infection (yeast, bacterial, or viral), symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants with a history of autoimmune disease such as systemic lupus erythematosus, celiac disease, autoimmune hepatitis, multiple sclerosis, exclusive of a history of thyroiditis, psoriasis, Sjrogen's, or inflammatory bowel disease.
* Pregnant and breastfeeding women are excluded from this study because pNGVL4aCRTE6E7L2 is a vaccine with unknown potential for teratogenic or abortifacient effects.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pNGVL4aCRTE6E7L2 DNA vaccine.
* Participants with a metal implant(s) at the site of injection or any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child.
* Syncopal episode within 12 months of screening.
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
* Individuals in which a skin-fold measurement of the cutaneous and subcutaneous tissue for all eligible injection sites (deltoid muscles with intact lymph drainage) exceeds 40 mm.
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art.
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical examination, previous EKG, and/or laboratory screening test.
* History of prior malignancy < 5 years; however individuals with completely resected basal cell or squamous cell carcinoma of the skin within this interval may be enrolled.
* Inability to understand or unwillingness to sign an informed consent document.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing dose limiting toxicities at each dosing level | 1 week
  The safety and tolerability of pNGVL4aCRTE6E7L2 DNA vaccine will be determined using the number of participants experiencing dose limiting toxicities at each dosing level.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Levinson, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Per our NCI grant resource sharing plan, this would include all coded data sets, including laboratory analyses of immune responses, as well as, if agreed to by participant, coded human specimens.
Time Frame: Immediately after publication of the study
Access Criteria: Sharing is governed by Johns Hopkins University Institutional Guidelines
URL: https://trp.cancer.gov/spores/abstracts/johnshopkins_gyn.htm